CLINICAL TRIAL: NCT01534338
Title: A Randomized Controlled Trial Testing the Effect of Mindfulness Practices Versus Sleep Education on Sleep and Inflammation Among Older Adults With Sleep Problems
Brief Title: Effect of Mindfulness Training on Sleep and Inflammation Among Older Adults With Sleep Problems
Acronym: MAPS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, David S. Black, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MH019925
Record Dates: First submitted 2012-02-09; First posted 2012-02-16 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Sleep Problems; Inflammation
Keywords: Sleep; inflammation; mindfulness; meditation; randomized controlled trial
MeSH Terms: conditions — Parasomnias; Inflammation | interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mindfulness Meditation (Experimental): The MAPs program is based on experiential training in mindfulness meditation offered at the UCLA Mindful Awareness Research Center (MARC). A certified UCLA instructor will provide didactic training in mindfulness meditation in a group-based setting. Participants will be guided through in-class meditation practices and will be assigned daily meditation homework. Active program components include sitting and walking somatosensory-focused meditation, audio-guided body scan meditation, and loving kindness meditation. Participants will attend weekly 2-hour classes for a total of 6 weeks and participants will monitor their sleep with a daily sleep diary. In addition to the MAPs training, sleep hygiene material will also be presented to match the sleep hygiene material in the sleep education condition.
  Interventions: Behavioral: Mindfulness Meditation
- Sleep Education (Active Comparator): The sleep education condition is founded on knowledge acquisition. In the sleep seminar condition, a trained health educator will provide didactic presentations on sleep, sleep hygiene, sleep problems, and potential solutions to sleep problems in a group-based setting. Active components of sleep education include increasing knowledge of sleep biology, identifying characteristics of healthy and unhealthy sleep, sleep problems, and self-monitoring of sleep behavior. Participants attend weekly 2-hour classes for a total of 6 weeks and participants will monitor their sleep with a daily sleep diary. The health education condition is comparable to MAPs in terms of time, attention, group support, and participant expectancy of a benefit in sleep parameters.
  Interventions: Behavioral: Sleep Education

INTERVENTIONS:
Behavioral: Mindfulness Meditation — Participants will attend weekly 2-hour classes for a total of 6 weeks and participants will monitor their sleep with a daily sleep diary.
  Arms: Mindfulness Meditation
Behavioral: Sleep Education — Participants will attend weekly 2-hour classes for a total of 6 weeks and participants will monitor their sleep with a daily sleep diary.
  Arms: Sleep Education

SUMMARY:
The primary aim of the study is to test the effect of mindfulness training on sleep parameters among older adults with insomnia symptoms

The secondary aims are to examine if changes in mindfulness meditation practice (daily log) and level of mindfulness (self-report) are associated with changes in sleep parameters, and to determine if mindfulness training is associated with in vitro biological markers of peripheral inflammation

ELIGIBILITY:
Inclusion Criteria:

* Men and women (all races and ethnicities) 55 years of age and older
* Have current problems sleeping
* Fluent in English
* Able to understand and provide signed informed consent
* Willing to be randomly assigned to treatment condition

Exclusion Criteria:

* Individuals currently undergoing major medical treatment such as surgery, radiation, or immunotherapy
* Individuals living outside of a 20 mile radius from the UCLA Medical Center
* Individuals with current substance dependence

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Sleep | Within 2 weeks post-intervention
  Primary sleep outcomes to be assessed include Daily sleep diary, Pittsburgh Sleep Quality Index, Fatigue Symptom Inventory, Insomnia Severity Index, and Pre-Sleep Arousal Scale

SECONDARY OUTCOMES:
Mindfulness | Within 2 weeks post-intervention
  Mindfulness will be assessed by self report with the Five Facet Mindfulness Questionnaire and a daily log of amount of mindfulness practice
Inflammatory Biology | Within 2 weeks post-intervention
  Pro-inflammatory cytokines and associated transcription markers will be assessed with in vitro assay of peripheral blood via venipuncture collected between 9am and 1130am

CONTACTS AND LOCATIONS:
Overall Officials: David S Black, M.P.H., Ph.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

REFERENCES:
- [Derived] Black DS, O'Reilly GA, Olmstead R, Breen EC, Irwin MR. Mindfulness meditation and improvement in sleep quality and daytime impairment among older adults with sleep disturbances: a randomized clinical trial. JAMA Intern Med. 2015 Apr;175(4):494-501. doi: 10.1001/jamainternmed.2014.8081. PMID 25686304